CLINICAL TRIAL: NCT03415724
Title: Comparison of Anesthetic Efficacy of Dexmedetomidine and Epinephrine in Combination With 2% Lidocaine for Inferior Alveolar Nerve Block in Patients With Irreversible Pulpitis: A Prospective, Double Blinded, Randomized Controlled Trial.
Brief Title: Comparison of Anesthetic Efficacy of Dexmedetomidine and Epinephrine With Lidocaine in Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Shreya singh
Record Dates: First submitted 2017-12-29; First posted 2018-01-30 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Irreversible Pulpitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1.8 ml Lignocaine plus adrenaline (Active Comparator): The study subjects will receive conventional inferior alveolar nerve block with 1.8 ml of 2% inj lignocaine with adrenaline 1:80000.
  Interventions: Procedure: Inferior alveolar nerve block
- 3.6 ml Lignocaine plus adrenaline (Active Comparator): The study subjects will receive conventional inferior alveolar nerve block with 3.6 ml of 2% inj lignocaine with adrenaline 1:80000.
  Interventions: Procedure: Inferior alveolar nerve block
- 1.8 ml Lignocaine plus dexmedetomidine (Active Comparator): conventional inferior alveolar nerve block with1.8 ml of injection lignocaine plus injection dexmedetomidiene 1micromol/ ml.
  Interventions: Procedure: Inferior alveolar nerve block
- 3.6 ml Lignocaine plus dexmedetomidine (Active Comparator): conventional inferior alveolar nerve block with3.6 ml of injection lignocaine plus injection dexmedetomidiene 1micromol/ ml.
  Interventions: Procedure: Inferior alveolar nerve block

INTERVENTIONS:
Procedure: Inferior alveolar nerve block — Inferior alveolar nerve block will be given to patients having irreversible pulpitis in mandibular molars

SUMMARY:
Aim of the study is to determine and compare the anaesthetic efficacy of dexmedetomidine and epinephrine in combination with 2% lidocaine for inferior nerve block in patients with irreversible pulpitis. Study will be conducted in Post Graduate Institute of Dental Sciences, Rohtak in department of Conservative Dentistry & Endodontics. Vital mature permanent mandibular molars with radiographically exposed dentinal caries and with signs of irreversible pulpitis will be included in the study. The patients will be randomly allocated into two control and two experimental groups and nerve block will be given according to standard protocol.

DETAILED DESCRIPTION:
AIMS AND OBJECTIVES:

To evaluate the efficacy of conventional inferior alveolar nerve block in mandibular molars with symptomatic irreversible pulpitis with injection dexmedetomidine plus injection lignocaine and compare it with injection lignocaine plus adrenaline.

MATERIALS AND METHODS - Study subjects will be recruited from OPD of Department of conservative dentistry and endodontics, PGIDS, Rohtak.

METHODOLOGY- Prior to treatment, a thorough clinical and radiological examination will be carried out and a thorough history will be taken.

Clinical procedure:

Mature mandibular permanent molars exhibiting deep caries involving pulp radiographically will be chosen for the study. The teeth will be evaluated by periapical radiographs, periodontal probing, percussion test, and vitality assessment with thermal test and electric pulp test; teeth determined to have irreversible pulpitis will be included and with reversible pulpitis will be excluded. All periapical radiographs will be exposed by using constant kVP, mA, and exposure time (70 KVP, 8 mA, and 0.8 sec.) with a Rinn paralleling device.

Study groups:

The subjects will be randomly assigned to 2 EXPERIMENTAL AND 2 CONTROL groups. CONTROL GROUP 1 - The study subjects will receive conventional inferior alveolar nerve block with 1.8 ml of 2% inj lignocaine with adrenaline 1:80000.

CONTROL GROUP 2 - The study subjects will receive conventional inferior alveolar nerve block with 3.6 ml of 2% inj lignocaine with adrenaline 1:80000.

EXPERIMENTAL GROUP 1 - conventional inferior alveolar nerve block with1.8 ml of injection lignocaine plus injection dexmedetomidine 1micromol/ ml.

EXPERIMENTAL GROUP 2 - conventional inferior alveolar nerve block with3.6 ml of injection lignocaine plus injection dexmedetomidine 1micromol/ ml.

* Patients will be explained the treatment procedure and use of pain scales.
* Patients will mark their pretreatment pain on a 170-mm HP VAS
* The area of injection will be dried by using sterile gauze, and topical anesthesia of 20% benzocaine (Mucopain; ICPA, Mumbai, India) will be applied by using sterile cotton-tip applicator for 60 seconds.
* The solution will be injected via a 5-mL disposable syringe (pricon, jodhpur, India) with a 24-gauge needle .
* The anterior border of the mandibular ramus will be palpated and coronoid notch located.
* The needle will be inserted on an imaginary line drawn from coronoid notch to the pterygomandibular raphe, 2 mm above the occlusal plane of mandibular molars.
* The barrel of the syringe will be in the opposite corner of the mouth, between the mandibular premolars.
* The needle will be inserted until bony resistance felt. After reaching the target area, aspiration will be performed, and the solution will be deposited with a rate of 1 ml/min. No anaesthetic solution will be deposited during needle insertion and placement.

Heft-parker visual analogue scale (Heft & Parker 1984), with 170-millimetre line marked with various terms describing the levels of pain, will be used. The millimetre marks will be removed from the scale, and the scale will be divided into 4 categories:

* 'no pain' corresponding to 0 mm;
* 'faint, weak or mild' pain corresponding to 1-54 mm;
* 'moderate' pain corresponding to 55-114 mm; and
* severe pain corresponding above 114 mm and included 'strong, intense and maximum possible' pain.

  * After 15 minutes, each patient will be asked whether his or her lip is numb.
  * If profound lip numbness is not recorded, the block will be considered unsuccessful, and the patients will be excluded from the study.
  * A conventional access opening will be initiated after isolation with a rubber dam. Patients will be instructed to raise their hand if any pain felt during the procedure.
  * In case of pain during the treatment, the procedure will be stopped, and patients will be asked to rate the pain on HP VAS.
  * The extent of access preparation and/or instrumentation will be recorded as
* within dentin,
* within pulpal space,
* and instrumentation of canals. • Success will be defined as no pain or weak/mild pain during endodontic access preparation and instrumentation

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age.
* Patient willing to participate in the study.
* Mature permanent mandibular first and second molars exhibiting signs of symptomatic irreversible pulpitis as assessed by history, cold and electric pulp tests.
* Absence of periapical lesions on radiographic examination.

Exclusion Criteria:

* Patient not ready to participate in the study voluntarily
* Clinical history or electrocardiographic evidence of heart block, Ischaemic heart disease
* Asthma, Sleep apnoea syndrome.
* Impaired liver, renal or mental function.
* Alcohol consumption in excess of 28 units per week.
* Chronic sedative and analgesic user and those having known allergy to study drugs
* Patients with severe periodontal disease.
* Patients unable to return for recall appointments
* Signs or symptoms of external /internal resorption, furcation or periapical radiolucency, swelling, or sinus tract.
* Negative response to cold and electric pulp tests.
* Antibiotic or analgesic intake within past 24 hours before treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
pain intensity | The root canal treatment will be completed in two sittings and the second sitting will be provided after 3-4 days.The time frame of the study is estimated to be about 6 months
  After giving inferior alveolar nerve block as per the standard protocol, conventional access opening will be initiated after isolation with a rubber dam. Patients will be instructed to raise their hand if any pain felt during the procedure and rate the pain on heft parker VAS scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No